CLINICAL TRIAL: NCT06303141
Title: Comparative Effects of Neuromuscular Training and Mobilization With Movement on Pain, Range of Motion, Function and Disability in Professional Athletes With Ankle Sprain
Brief Title: Comparative Effects of Neuromuscular Training and Mobilization With Movement in Professional Athletes With Ankle Sprain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LUC/CPGS/PGS/20230405/001
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Ankle Injuries; Musculoskeletal Manipulations
Keywords: NEUROMUSCULAR TRAINING; MOBILIZATION WITH MOVEMENT; Professional Athletes; Ankle Sprain
MeSH Terms: conditions — Ankle Injuries | interventions — Movement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the assessor who take the reading is blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Closed Chain Exercises (Other): Group A, serving as the control group, will undergo a structured rehabilitation regimen comprising closed chain exercises, icing, and bracing. The exercise component will focus on enhancing proprioception and strengthening the ankle joint. Participants will perform exercises including open eyes and closed eyes across arm movements for three sets lasting 60 seconds each, lateral step down exercises for three sets of 6-12 repetitions, semi-squat exercises for three sets of 6-12 repetitions, and Thera-band isometric exercises for three sets of 10-15 seconds each. These exercises are designed to promote ankle stability, improve range of motion, and enhance muscle strength. Additionally, icing and bracing will be utilized to reduce inflammation and provide external support to the injured ankle.
  Interventions: Other: Closed Chain exercises
- Neuromuscular training (Experimental): Group B, designated as the experimental group, will undergo a comprehensive rehabilitation protocol combining neuromuscular training with closed chain exercises, icing, and bracing. The exercise regimen will target proprioception, neuromuscular control, and ankle stability. Participants will engage in a series of exercises including single leg raises for three sets lasting 30 seconds each, ankle eversion/inversion exercises for three sets of 25 repetitions, double hopping in place then out of place for three sets of 30 seconds, reaching exercises with feet and hands for three sets lasting 30-60 seconds each, and wobble board exercises for three sets lasting 30-60 seconds each. These exercises are aimed at improving balance, coordination, and muscle strength around the ankle joint. The addition of neuromuscular training enhances the proprioceptive feedback and control, which is crucial for injury prevention and functional recovery in athletes with ankle sprains.
  Interventions: Other: Neuromuscular Training
- Mobilization with movement (Experimental): Group C, designated as an experimental group, will undergo a unique intervention combining mobilization with movement techniques, closed chain exercises, icing, and bracing. The focus of this intervention is to address joint dysfunctions and pain modulation while improving range of motion (ROM) in athletes with ankle sprains. Participants will receive joint mobilization with movement techniques, following the Mulligan approach, aimed at restoring normal joint mechanics and function. The protocol will involve three sets of six oscillations or glides each, targeting specific joint restrictions and impairments associated with ankle sprains. By integrating manual therapy with exercise and adjunct modalities like icing and bracing, this comprehensive approach aims to optimize joint function, reduce pain, and enhance overall rehabilitation outcomes in professional athletes with ankle injuries.
  Interventions: Other: Mobilization with Movement

INTERVENTIONS:
Other: Closed Chain exercises — Open eyes and closed eyes across arm" (3 sets x 60 sec) Lateral step down (3 sets x 6-12 reps) Semi-Squat Exercise (3sets x 6-12 reps) Thera-band isometric (3 sets x 10 -15sec each)
  Arms: Closed Chain Exercises
Other: Neuromuscular Training — Neuromuscular Training Exercise:
  * Single Leg Raise (3 sec x 30sec each)
  * Ankle eversion/inversion (3 sets x 25 reps)
  * Double Hopping in place then out of place (3 sets 30 sec)
  * Reach with feet (3 sets x 30-60 sec each)
  * Reach with hands (3 sets x 30-60 sec each)
  * Wobble board Exercise (3sets x 30-60sec each
  Arms: Neuromuscular training
Other: Mobilization with Movement — Joint mobilization with movement (by Mulligan) refers to manual therapy techniques that are used to modulate pain and treat joint dysfunctions that limit the range of motion (ROM).
  (3 sets x 6 oscillation/glide each)
  Arms: Mobilization with movement

SUMMARY:
The study aims to compare the effects of neuromuscular training and mobilization with movement on pain, range of motion, function, and disability in professional athletes with ankle sprain. Neuromuscular training focuses on improving neuromuscular control and stability, while mobilization with movement aims to restore joint mobility and function. By investigating the outcomes of these two interventions, the study seeks to provide insights into their effectiveness for managing ankle sprains in professional athletes.

DETAILED DESCRIPTION:
The comparative study on the effects of neuromuscular training and mobilization with movement on pain, range of motion, function, and disability in professional athletes with ankle sprain is designed to address the efficacy of these two interventions in managing ankle injuries among athletes. An ankle sprain is a common injury in sports, often resulting in pain, limited range of motion, functional impairment, and disability. Therefore, identifying the most effective treatment approaches is essential for promoting athletes' recovery and minimizing the impact of ankle sprains on their performance.

Neuromuscular training is a structured exercise program aimed at improving neuromuscular control, proprioception, balance, and strength around the ankle joint. It typically involves exercises targeting the muscles and ligaments involved in ankle stability, such as balance training, proprioceptive exercises, strength training, and functional rehabilitation exercises. The goal of neuromuscular training is to enhance joint stability, reduce the risk of re-injury, and improve functional outcomes in athletes with ankle sprains.

On the other hand, mobilization with movement is a manual therapy technique used to restore joint mobility and function through specific movements or mobilizations. This approach involves applying controlled and graded movements to the affected ankle joint while simultaneously mobilizing the surrounding soft tissues. Mobilization with movement aims to reduce pain, improve joint mobility, and restore normal movement patterns by addressing restrictions in joint mobility, muscle tightness, and soft tissue adhesions.

The comparative study will involve professional athletes who have sustained ankle sprains during sports participation. Participants will be randomly assigned to either the neuromuscular training group or the mobilization with movement group. Both groups will undergo a structured intervention program tailored to their respective treatment approach.

The neuromuscular training program will consist of a series of progressive exercises targeting ankle stability, balance, strength, and proprioception. These exercises may include single-leg balance exercises, resistance training using bands or weights, agility drills, plyometric exercises, and functional activities relevant to the athlete's sport.

Meanwhile, the mobilization with movement intervention will involve manual therapy techniques administered by a qualified physiotherapist or sports therapist. These techniques may include joint mobilizations, soft tissue mobilizations, and specific movement patterns designed to restore normal joint mechanics and improve ankle function.

Outcome measures will include pain levels, range of motion (assessed using goniometry), functional status (evaluated using standardized outcome measures such as the Foot and Ankle Ability Measure), and disability scores (measured using validated scales such as the Disability Rating Index). These measures will be assessed at baseline, post-intervention, and follow-up time points to evaluate the effectiveness of each intervention in improving ankle sprain outcomes.

The study's findings will provide valuable insights into the comparative effectiveness of neuromuscular training and mobilization with movement in professional athletes with ankle sprains. By identifying the most beneficial treatment approach, the study aims to optimize rehabilitation strategies for ankle injuries in athletes, ultimately supporting their return to sport and minimizing the risk of re-injury.

ELIGIBILITY:
Inclusion Criteria:

* • Athletes will be included:

  * Rackets player,
  * Basketball players
  * Runners
  * Foot-ballers players
  * Soccer players,
  * and Volley-ball players
  * Gender: both male and female
  * Age: 18 to 35 years old
  * Training: 15-20/ week
  * Sustained an ankle sprain grade II and III
  * With no Functional Ankle Instability (Greek version of the Identification functional ankle instability questionnaire IdFAI, score < 10) will be used in order to identify athletes with FAI

Exclusion Criteria:

* • Any vestibular or balance disorders (1)

  * History of surgery and trauma of a lower limb since last 6 months
  * Athletes with pain related to calf muscles and achillies tendon
  * Co-morbidities: Diabetes, Hypertension, etc

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale for Pain | 4 weeks
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an elevenpoint numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Goniometer for Range of Motion | 4 weeks
  A goniometer is a device that measures an angle or permits the rotation of an object to a definite position
Star balance excursion test for Balance | 4 weeks
  The Star Excursion Balance Test is a reliable measure and a valid dynamic test to predict risk of lower extremity injury, to identify dynamic balance deficits in patients with lower extremity conditions, and to be responsive to training programs in healthy participants and those with lower extremity conditions.
Foot and ankle ability Measure for Functional Performance | 4 weeks
  The FAAM is a self-report measure that assesses physical function of individuals with lower leg, foot, and ankle musculoskeletal disorders. 2) Sports subscale of 8 items. For each subscale patients are asked to answer each question with a single response that most clearly describes their condition within the past week.
Cumberland Ankle Instability | 4 weeks
  The Cumberland Ankle Instability Tool (CAIT) is a self-report questionnaire used to assess the severity of chronic ankle instability (CAI). It consists of nine items designed to evaluate functional ankle instability, including symptoms of giving way, recurrent sprains, and perceived ankle function during daily activities. Each item is scored on a 0 to 30 scale, with higher scores indicating better ankle stability

SECONDARY OUTCOMES:
Agility T-test | 4 weeks
  The Agility T-Test is a widely used physical performance test designed to assess an individual's agility, speed, and quickness. It involves a series of directional changes and sprints around cones or markers arranged in a T-shape. The test measures the time taken by the individual to complete the course accurately. It requires rapid acceleration, deceleration, and changes of direction in multiple planes of movement, making it a comprehensive assessment of agility and dynamic balance. The Agility T-Test is commonly used in sports performance testing, fitness evaluations, and rehabilitation settings to assess an individual's agility and athletic ability.
Speed (20m sprint test) | 4 weeks
  The 20-meter sprint test is a commonly used measure of an individual's speed and acceleration. In this test, the participant is required to sprint as fast as possible over a distance of 20 meters from a standing start. The time taken to complete the sprint is recorded using timing gates or a stopwatch, providing a measure of the participant's sprinting speed.
  The 20-meter sprint test is often used in sports performance assessments, fitness testing, and research studies to evaluate an individual's anaerobic power and speed capabilities. It is particularly relevant for athletes competing in sports that require short bursts of maximal effort, such as sprinting, soccer, basketball, and rugby

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Gul Memon, PhD Scholar, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No